CLINICAL TRIAL: NCT06841172
Title: Continuation of First-line Therapy With Radiotherapy for Oligoprogression Versus Early Switch to Second-line Therapy in Oligoprogressive Hepatocellular Carcinoma (CROSS): a Multi-center, Randomized, Controlled, Open-label, Phase Ⅲ Trial
Brief Title: Continuation of First-line Therapy With Radiotherapy Versus Early Switch to Second-line Therapy in Oligoprogressive HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-025-02
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: OligoProgressive Metastatic Disease; Hepatocellular Carcinoma (HCC); Radiotherapy; Systemic Therapy
Keywords: oligoprogressive; HCC; radiotherapy; first-line systemic therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy group (Experimental): Patients will continue their current first-line systemic treatment, which may include, but is not limited to, combinations such as atezolizumab plus bevacizumab, tremelimumab plus durvalumab, or monotherapies such as lenvatinib, sorafenib, tislelizumab, durvalumab, or pembrolizumab, at the discretion of the treating physician. All oligoprogressive lesions will receive radiotherapy. Radiotherapy Techniques: 3D-CRT, IMRT, IGRT. Radiation dose and fractionation: radiation dose will be biologically effective dose (BED) ≥60 Gy, adjusted based on tumor location and size. For intrahepatic oligoprogressive lesions, eligibility for radiotherapy is determined by multidisciplinary team (MDT) consultation, and patients must meet the following criteria
  1. Residual normal liver volume ≥700 mL
  2. D ≥ 700 cc ≤ 23 Gy (for Child-Pugh B patients) If oligoprogression recurs after ≥3 months, additional radiotherapy will be administered in addition to continuation of current first-line systemic therapy.
  Interventions: Radiation: radiotherapy; Drug: Systemic therapy (Continuation of current first-line systemic therapy)
- Control (Active Comparator): For patients who received sorafenib as FLST, regorafenib will be the preferred second-line option. For patients who received other FLST regimens, the SLST selection will be determined through an MDT discussion led by the treating physician based on the patient's overall condition, prior therapies, drug indications, and potential adverse effects, ensuring an individualized treatment approach. The specific dosing regimen, administration frequency, and dose adjustments will strictly follow the same prescribing information for each drug.
  Interventions: Drug: Systemic therapy (Early switch to second-line systemic therapy)

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy (Biologically Equivalent Dose [BED]≥60Gy)
  Other Names: RT
  Arms: Radiotherapy group
Drug: Systemic therapy (Continuation of current first-line systemic therapy) — Continuation of current first-line systemic therapy, which may include, but is not limited to, combinations such as atezolizumab plus bevacizumab, tremelimumab plus durvalumab, or monotherapies such as lenvatinib, sorafenib, tislelizumab, durvalumab, or pembrolizumab, at the discretion of the treating physician.
  Other Names: c-FLST
  Arms: Radiotherapy group
Drug: Systemic therapy (Early switch to second-line systemic therapy) — For patients who received sorafenib as FLST, regorafenib will be the preferred second-line option. For patients who received other FLST regimens, the SLST selection will be determined through an MDT discussion led by the treating physician based on the patient's overall condition, prior therapies, drug indications, and potential adverse effects, ensuring an individualized treatment approach. The specific dosing regimen, administration frequency, and dose adjustments will strictly follow the same prescribing information for each drug.
  Other Names: s-SLST
  Arms: Control

SUMMARY:
This multicenter, prospective, randomized, controlled, open-label, two-arm Phase III clinical trial is designed to evaluate whether adding radiotherapy to oligoprogressive lesions while continuing first-line systemic therapy at the time of oligoprogression can effectively prolong progression-free survival compared to early switching to second-line systemic therapy in oligoprogressive hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is often diagnosed at an advanced stage due to its aggressive nature and lack of early symptoms, making most patients ineligible for curative treatment. In recent years, novel therapeutic approaches, including targeted therapy, immunotherapy and combination regimens, have improved systemic treatment outcomes for advanced HCC, thereby increasing patient survival. However, the objective response rate of first-line systemic treatments remains limited at approximately 20-35%, and most patients inevitably develop resistance and disease progression during treatment.

For patients undergoing first-line systemic therapy (FLST) who develop oligoprogression - defined as the progression of a limited number of lesions during systemic treatment - the standard approach is typically to move to second-line systemic therapy (SLST). However, available SLST options remain limited, with median progression-free survival (PFS) of only 2.6-3.1 months, underscoring the urgent need for optimized treatment strategies.

The investigators hypothesize that administering local radiotherapy to oligoprogressive lesions while continuing current FLST - provided it remains effective for non-progressing disease - could delay the need for SLST and potentially improve both PFS and OS. This treatment approach has been validated in prospective studies in other malignancies. In addition, our recent multicenter retrospective study published in the Red Journal demonstrated that maintaining FLST in combination with radiotherapy for oligoprogressive lesions significantly prolonged PFS in patients with HCC.

Based on these findings, this study aims to conduct a prospective, randomized, controlled Phase III clinical trial in patients with oligoprogressive HCC following FLST. The trial will evaluate whether adding radiotherapy to oligoprogressive lesions while continuing current FLST provides clinical benefit compared to early transition to SLST.

The primary endpoint of this trial is PFS. The secondary endpoints include OS, objective response rate (ORR), disease control rate (DCR), duration of response (DOR), and safety (assessed according to CTCAE 5.0).

This trial will enroll patients with HCC who experience oligoprogression while receiving FLST, provided they have received at least three months of FLST prior to oligoprogression. Patients will be randomized 1:1 to one of two cohorts:

Cohort 1: Radiotherapy targeting oligoprogressive lesions while continuing current FLST.

Cohort 2: Early transition to SLST. In addition, exploratory objectives include the collection and analysis of circulating tumor DNA (ctDNA) to assess dynamic changes at baseline (time of oligoprogression), at first follow-up after radiotherapy, and at subsequent disease progression. A subset of participants will also undergo biopsies of both primary tumors and progressive lesions at baseline (oligoprogression) and at subsequent progression to further investigate molecular and genomic changes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histological or cytological confirmation of primary hepatocellular carcinoma (HCC), or diagnosis based on the Clinical Diagnosis and Treatment Guidelines for Primary Liver Cancer (2024 edition) issued by the National Health Commission of the People's Republic of China.
* 2. BCLC stage C at the time of first-line systemic treatment.
* 3. Oligoprogression must be confirmed by imaging or histopathology during first-line systemic therapy (FLST). The number of oligoprogressive lesions is limited to 1-5, involving no more than 1-3 organs or systems. These lesions may represent either new metastatic sites or progression of pre-existing lesions. In addition, they must fit one of the two classifications defined in the ESTRO-EORTC consensus on oligometastases: repeat oligoprogression or induced oligoprogression. Oligoprogression may occur within intrahepatic lesions. In the case of lymph node progression, each lymphatic drainage region is considered a separate lesion. For example, the para-aortic lymph nodes (number 16a and number 16b) are each counted as separate lymph node regions.
* 4. Patients must have experienced oligoprogression while receiving their current FLST and must not have previously received any other FLST that resulted in disease progression. Additionally, the current FLST must have maintained disease stability (SD) for at least three months prior to the occurrence of oligoprogression. Furthermore, the expected survival time must be ≥6 months.
* 5. Oligoprogressive lesions must be eligible for radiotherapy and should have at least one measurable lesion that meets RECIST v1.1 criteria; Bone metastases without soft tissue formation are eligible but are considered non-measurable lesions; Bone metastases with soft tissue formation that meet RECIST v1.1 measurable criteria are considered measurable lesions.
* 6. Liver function must be assessed as Child-Pugh score ≤7 points.
* 7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-1.
* 8. Participants must be able to understand and voluntarily sign a written informed consent prior to the initiation of any study-specific procedures and must agree to comply with the treatment and follow-up requirements of the study.
* 9. Male or female patients between 18 and 75 years of age.
* 10. Availability of tumor and blood samples for biomarker assessment.

Exclusion Criteria:

* 1. Patients who received FLST as adjuvant treatment after curative surgery for HCC.
* 2. Tumor progression occurring within 3 months after initiation of FLST.
* 3. Patients with combined hepatocellular-cholangiocarcinoma (cHCC-CC)
* 4. History of grade ≥3 serious adverse events due to FLST.
* 5. Presence of brain, peritoneal or omental metastases with bleeding after FLST.
* 6. Previous radiation therapy to the site of the oligoprogressive lesion.
* 7. Active untreated hepatitis B, defined as HBsAg positive with HBV DNA levels above the upper limit of normal in the participating center's laboratory.
* 8. Oligoprogressive lesions not amenable to radiotherapy.
* 9. Alpha-fetoprotein (AFP) level ≥10,000 ng/mL at the time of oligoprogression.
* 10. Diagnosis of malignancy other than liver cancer within 3 years prior to enrollment (excluding curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, and/or carcinoma in situ).
* 11. Currently participating in any interventional clinical research treatment or having received any other investigational drug or investigational device therapy within the last 4 weeks prior to enrollment.
* 12. Presence of autoimmune disease or other conditions requiring long-term steroid use.
* 13. Severe impairment of the heart, lungs, kidneys, or other vital organs, active infections (other than viral hepatitis), or other serious comorbidities that render the patient unable to tolerate treatment.
* 14. known or suspected allergy to any study drug or to any drug related to this study.
* 15. History of organ transplantation
* 16. Pregnant or breastfeeding women
* 17. Any other factor that the investigator believes may affect the enrollment of patients or the evaluation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  The time between enrollment and disease progression or death for patients in the intent-to-treat population, whichever occurred first; for those who did not progress at the time of withdrawal from the study or whose time to disease progression was not recorded, the date of the last visit was used as the endpoint date.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Defined as the time from initiation of treatment to death from any cause.
Adverse event incidence (Safety) | 2 years
  Treatment-related adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE 5.0).
Objective response rate (ORR) | 2 years
  Defined as the proportion of patients whose tumor size decreases (partial response) or disappears (complete response) after radiation based on RECIST 1.1.
Disease control rate (DCR) | 2 years
  Defined as the proportion of patients whose tumor size decreases (partial response), disappears (complete response), or is stable after radiation based on RECIST 1.1.
Duration of response (DOR) | 2 years
  Defined as the time in patients whose tumor size decreases (partial response), disappears (complete response), or is stable after radiation based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Jinan, Shandong 0531, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leng B, Wang H, Ge Y, Sun X, Dong P, Dong X, Duan X, Wang Q, Xia Y, Ding L, Dai H, Liu T, Shi F, Zhang X, Yue J. Maintaining First-Line Therapy Plus Radiation Therapy May Prolong Progression-Free Survival and Delay Second-Line Therapy for Oligoprogressive Hepatocellular Carcinoma. Int J Radiat Oncol Biol Phys. 2025 Jun 1;122(2):325-338. doi: 10.1016/j.ijrobp.2024.12.039. Epub 2025 Jan 15. PMID 39824367
- [Background] Choi SH, Lee BM, Kim J, Kim DY, Seong J. Efficacy of stereotactic ablative radiotherapy in patients with oligometastatic hepatocellular carcinoma: A phase II study. J Hepatol. 2024 Jul;81(1):84-92. doi: 10.1016/j.jhep.2024.03.003. Epub 2024 Mar 11. PMID 38467379
- [Background] Doyle E, Killean AJ, Harrow S, Phillips ID. Systematic review of the efficacy of stereotactic ablative radiotherapy for oligoprogressive disease in metastatic cancer. Radiother Oncol. 2024 Jul;196:110288. doi: 10.1016/j.radonc.2024.110288. Epub 2024 Apr 20. PMID 38648995
- [Background] Tan VS, Padayachee J, Rodrigues GB, Navarro I, Shah PS, Palma DA, Barry A, Fazelzad R, Raphael J, Helou J. Stereotactic ablative radiotherapy for oligoprogressive solid tumours: A systematic review and meta-analysis. Radiother Oncol. 2024 Nov;200:110505. doi: 10.1016/j.radonc.2024.110505. Epub 2024 Aug 26. PMID 39197501
- [Background] Wang Q, Yu J, Sun X, Li J, Cao S, Han Y, Wang H, Yang Z, Li J, Hu C, Zhang Y, Jin L. Sequencing of systemic therapy in unresectable hepatocellular carcinoma: A systematic review and Bayesian network meta-analysis of randomized clinical trials. Crit Rev Oncol Hematol. 2024 Dec;204:104522. doi: 10.1016/j.critrevonc.2024.104522. Epub 2024 Sep 26. PMID 39332750
- [Background] Cappuyns S, Corbett V, Yarchoan M, Finn RS, Llovet JM. Critical Appraisal of Guideline Recommendations on Systemic Therapies for Advanced Hepatocellular Carcinoma: A Review. JAMA Oncol. 2024 Mar 1;10(3):395-404. doi: 10.1001/jamaoncol.2023.2677. PMID 37535375
- [Background] Llovet JM, Castet F, Heikenwalder M, Maini MK, Mazzaferro V, Pinato DJ, Pikarsky E, Zhu AX, Finn RS. Immunotherapies for hepatocellular carcinoma. Nat Rev Clin Oncol. 2022 Mar;19(3):151-172. doi: 10.1038/s41571-021-00573-2. Epub 2021 Nov 11. PMID 34764464
- [Background] Quail DF, Joyce JA. Microenvironmental regulation of tumor progression and metastasis. Nat Med. 2013 Nov;19(11):1423-37. doi: 10.1038/nm.3394. PMID 24202395